CLINICAL TRIAL: NCT06832475
Title: Effects of Class II Elastics During Treatment with Clear Aligners Vs Fixed Appliance: a Randomized Clinical Trial
Brief Title: Comparing the Impact of Rubber Bands on Teeth Straightening with Clear Aligners Versus Traditional Braces: a Clinical Study
Acronym: Class II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppina Laganà, EFFECTS OF CLASS II ELASTICS DURING TREATMENT WITH CLEAR ALIGNERS VS FIXED APPLIANCE: A RANDOMIZED CLINICAL TRIAL, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethical Commitee n. 24/23
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Class II Malocclusion; IMPA Angle
MeSH Terms: conditions — Overbite | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: randomized clinical trial, blinded about the type of treatment
Who Masked: Participant
Masking Description: the partecipants didn't know which type of treatment they will have
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Class II malocclusion with clear aligners (Experimental): For the groupteated with Clear Aligners (CA), the treatment provided the application of Invisalign clear aligner system and the absence of any other auxiliaries apart from Invisalign optimized attachments. Each subject was instructed to wear aligners for 22 hours per day, except during meals and oral hygiene procedures and to replace aligners once a week, always the same day of the week. Every six stages the clinician personally checked the good aligner fitting, the position of the attachments and the patient collaboration.
  Interventions: Device: clear aligners and elastics; Device: class 2 elastics
- Class II malocclusion with fixed appliance and elastics (Experimental): For the group treated with Fixed Appliance (FA), the straight wire treatment included an aligning and leveling phase, achieved by using Nickel-Titanium arches (0.016/0.019 × 0.025 arc sequence) and a phase with heavier stainless steel rectangular arches (0.019 × 0.025); during this last treatment phase patients were instructed to use Class II elastics for at least 16 h/day.
  Pre- (T0) and post-treatment (T1) lateral cephalogram were collected from all selected patients. Treatment time was an average of 18 months (T1-T0=18 months).
  Interventions: Device: class 2 elastics

INTERVENTIONS:
Device: clear aligners and elastics — For the Fixed Appliance group, the straight wire treatment included an aligning and leveling phase, achieved by using Nickel-Titanium arches (0.016/0.019 × 0.025 arc sequence) and a phase with heavier stainless steel rectangular arches (0.019 × 0.025); during this last treatment phase patients were instructed to use Class II elastics for at least 16 h/day.
  Pre- (T0) and post-treatment (T1) lateral cephalogram were collected from all selected patients. Treatment time was an average of 18 months (T1-T0=18 months).
  Other Names: fixed appliance and elastics
  Arms: Class II malocclusion with clear aligners
Device: class 2 elastics — Class II malocclusion is the most common malocclusion, and it is one of the main reasons for people to undergo orthodontic treatment. This alteration is characterized by an improper relationship between the maxillary and mandibular arches because of skeletal or dental discrepancies or a combination of both . The treatment protocols may considerably vary depending on professional skills, malocclusion severity and patient compliance . Among all the well-known techniques, it is important to mention the Class II elastics , used to camouflage mild skeletal Class II or to treat mild to moderate Class II occlusal relationship.
  During the correction of Class II malocclusions by means of inter-arch elastics, special attention should be paid to the position of the lower incisors.

SUMMARY:
Aim: To analyze the inclination of lower incisors in patients with Class II malocclusion treated with elastics and clear aligners compared to a group wearing the same elastics and fixed appliance. A sample of 40 patients (19M and 21F), mean age 15.4±1.8 years, was randomly divided in two groups: Clear aligner group (CA), Fixed appliance group (FA). The subjects were selected according to inclusion criteria: full permanent dentition (excluding third molars), Class II molar relationship (2,5-4 mm), no history of orthodontic treatment.

DETAILED DESCRIPTION:
Trial design: Prospective two-arms parallel group randomized clinical trial with 1:1 allocation ratio.

Materials and Methods: A sample of 40 patients (19M and 21F), mean age 15.4±1.8 years, was collected from the Department of Orthodontics at Policlinico "Tor Vergata" of Rome, and it was randomly divided in two groups: Clear aligner group (CA), Fixed appliance group (FA). The subjects were selected according to inclusion criteria: full permanent dentition (excluding third molars), Class II molar relationship (2,5-4 mm), no history of orthodontic treatment. Results: In the short term (T1-T0=18 months), the analysis of the results showed no statistically significant changes in all evaluated parameters. Therefore, there is no statistically significant change in the inclination of the lower incisors between the two groups.

Conclusions: The use of Class II elastics in CA group showed a better control of the lower incisors' inclination, compared to the FA group, even if the difference is not significant.

Trial registration: ClinicalTrials.gov (registration number: ..........)

ELIGIBILITY:
Inclusion Criteria:

* full permanent dentition (excluding third molars), Class II molar relationship (2,5-4 mm), no or moderate crowding (0- 3 mm) no history of orthodontic treatment.

Exclusion Criteria:

* not completed permanent dentition, skeletal Class II or dental Class II more than 4 mm, crowding more than 3 mm, subjects already treated with iother orthodontic appliances.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Comparison between two different devices to solve class II dental malocclusion | From enrollment to the end of treatment at 18 months
  A sample of 40 patients (19M and 21F), mean age 15.4±1.8 years was collected from the Department of Orthodontics at Policlinico "Tor Vergata" of Rome, from September 2023 to June 2024. The sample was randomly divided in two groups: FA group (Fixed Appliance), consisted of 20 patients (9 M, 11F) treated by straight-wire fixed appliance and Class II elastics: CA group (Clear Aligners), consisted of 20 patients (9M, 11F) treated by Comprehensive Package Invisalign® system and Class II elastics. For both FA and CA groups, the inclusion criteria were the following: full permanent dentition (excluding third molars), Class II molar relationship (2,5-4 mm), no or moderate crowding (0- 3 mm) no history of orthodontic treatment.
  Pre- (T0) and post-treatment (T1) lateral cephalogram were collected from all selected patients. Treatment time was an average of 18 months (T1-T0=18 months).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tor Vergata, Rome, Rome, Italy

REFERENCES:
- [Derived] Lagana G, Malara A, Lione R, Bollero P, Cozza P. Effects of Class II elastics on lower incisors during treatment with clear aligners vs. fixed appliance: a randomized clinical trial. Front Dent Med. 2025 Jul 10;6:1613037. doi: 10.3389/fdmed.2025.1613037. eCollection 2025. PMID 40708614